CLINICAL TRIAL: NCT06724861
Title: Sensory Rehabilitation in CIPN
Brief Title: Sensory Rehabilitation in Chemo Induced Peripheral Neuropathy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Collaborators: Zefat Academic College (Other)
Responsible Party: Principal Investigator, Rotem Merose, MD, Assaf-Harofeh Medical Center
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CIPN - RCT
Record Dates: First submitted 2024-11-21; First posted 2024-12-09 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: CIPN - Chemotherapy-Induced Peripheral Neuropathy; Age Over 18; Chemotherapy-induced Peripheral Neuropathy
Keywords: Neuropathic pain; Chemo Induced Peripheral Neuropathy (CIPN); Sensory rehabilitation; Explicit Sensory Retraining; Lower extremity
MeSH Terms: conditions — Neuralgia

STUDY DESIGN:
Intervention Model Description: A Randomized Controlled Trial will be conducted in a within-subject cross-over design (AB BA). Full assessments will be conducted at baseline, after last treatment session. A short assessment will be conducted at the beginning of all sessions. The early intervention group (AB) will be assessed at one-month follow-up in addition. The later intervention group (BA) will be assessed at baseline, and after a month before treatment commences and immediately after last treatment
Who Masked: Investigator, Outcomes Assessor
Masking Description: The outcome assessor will not be aware of randomization and allocation. Primary investigator and statistician will receive data ready for analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- AB - early experimental treatment, later control usual care (Other): AB - early experimental treatment, later control usual care
  Interventions: Other: Explicit Sensory Retraining for the lower extremities; Other: no treatment
- BA - early control usual care, later experimental treatment (Other): BA - early control usual care, later experimental treatment
  Interventions: Other: Explicit Sensory Retraining for the lower extremities; Other: no treatment

INTERVENTIONS:
Other: Explicit Sensory Retraining for the lower extremities — Sensory retraining of detection, discrimination, quantification of a stimuli and recognition of stimuli and objects with the leg and mainly with the foot. Top-down awareness of bottom-up sensory experience in the treatment session and in everyday life.
Other: no treatment — Usual care

SUMMARY:
This study is a cross-over RCT evaluating the effectiveness of 3 sessions a week apart of explicit sensory retraining to the lower extremities in individuals with CIPN versus usual care. The primary outcome measures are TNAS for subjective symptoms, VAS for pain and TUG for mobility. Additional outcome measures are FABS for balance, sensory assessments - monofilaments for touch threshold, LEPT for proprioception, a home exercise log and a satisfaction questionnaire.

DETAILED DESCRIPTION:
Chemotherapy Induced Peripheral Neuropathy (CIPN) is a neurological complication of chemotherapy, affecting between 50%-90% of the patients: up to 68% within the first month after chemotherapy, 60% after 3 months, and 30% after 6 months.

Neuropathic symptoms can persist in 11% to more than 80% of individuals post chemotherapy at one to three years following treatment and around 50% even after 5 years and more.

CIPN is associated with lower self-reported physical function and Quality of Life (QoL).

The clinical picture is typically sensory, with involvement of large and small sensory fibers. Motor and autonomic involvement is less frequent.

Damage to sensory nerve fibers is typically symmetrical. Sensory loss in a 'glove and stocking type' distribution leads to 'minus' symptoms (loss of function) including numbness in hands and feet, impaired perception of light touch, hypoalgesia and impaired proprioception, temperature and vibration sensation. Paradoxically, 'plus' features (gain of function) such as paresthesia (tingling like pins and needles), dysesthesia, allodynia and hyperalgesia appear simultaneously. CIPN can be functionally debilitating including impaired balance, walking slower and shorter steps and increased falls.

Active, explicit sensory rehabilitation is efficient in promoting sensation and function in individuals with neurological conditions, such as stroke and multiple sclerosis. To the best of our knowledge although CIPN is primarily a sensory deficit there is no treatment aimed at this aspect. We aim to conduct a pilot study to explore the feasibility and clinical benefit of an active, explicit sensory rehabilitation protocol for the lower limb in individuals with chronic CIPN.

This study is a cross-over RCT evaluating the effectiveness of 3 sessions a week apart of explicit sensory retraining to the lower extremities in individuals with CIPN versus usual care. The primary outcome measures are TNAS for subjective symptoms, VAS for pain and TUG for mobility. Additional outcome measures are FABS for balance, sensory assessments - monofilaments for touch threshold, LEPT for proprioception, a home exercise log and a satisfaction questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* CIPN by self-report (present or absent) > 3 months after last chemotherapy treatment
* age > 18.

Exclusion Criteria:

* Pre-chemotherapy neuropathy/ sensory impairment
* recurrent falls prior to chemotherapy (more than 2 per year)
* CNS involvement
* not ambulatory before chemotherapy
* Hebrew proficiency not meeting questionnaires' needs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2024-12-11 (Estimated); Primary Completion 2024-12-11 (Estimated); Study Completion 2026-12-11 (Estimated)

PRIMARY OUTCOMES:
Patient self-Report Outcome Measure - Treatment-Induced Neuropathy Assessment Scale (TNAS) | from randomization 3 months maximum
  TNAS -Treatment-Induced Neuropathy Assessment Scale: patient-reported outcome measure of presence and severity of CIPN. Nine 0-10 question scale. score 0-90. A higher score is for higher CIPN symptom severity.
Functional - Balance and mobility outcome measure - Timed Up and Go test (TUG) | from randomization to maximum 3 months followup
  TUG -Timed Up and Go: Balance and mobility assessment. Serves as a fall prediction screening test. Measures time taken to raise from a chair walking 3 meters and re-sit.
Pain intensity: VAS - 0-100 mm visual scale | from randomization to maximum 3 months
  Pain intensity: VAS - 0-100 mm visual scale: self-reporting pain assessment from no pain to worst pain possible. We will ask for current pain and the worst pain during the last week

SECONDARY OUTCOMES:
Tactile function assessment - Semmes Weinstein Monofilaments (SWM) | from randomization to maximum 3 months followup
  Sensory threshold at the foot, as measured by Semmes Weinstein filaments.
FABS - Fullerton Advanced Balance Scale | from randomization to maximum 3 months
  FABS - Fullerton Advanced Balance Scale: high function balance test - consisting of 10 activities in both static and dynamic phases; 10-40, higher scores are better.
Proprioception of lower extremity: Lower Extremity Position Test (LEPT) | from randomization to maximum 3 months followup
  Proprioception of lower extremity as measured by Lower Extremity Position Test (LEPT).

OTHER OUTCOMES:
Home exercise log | 1 minutes writing daily at home
  Amount of home exercise per minutes per day
Participant satisfaction questionnaire | 5 minutes, at final assessment session only
  Participant satisfaction questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Asaph-Harofe Shamir Medical Center, Rishon LeZiyyon, Israel

IPD SHARING:
Plan to Share IPD: Undecided